CLINICAL TRIAL: NCT07158073
Title: The Effect of Oxygen Reserve Index Guided Oxygen Titration on Oxidative Stress in Rhinoplasty Surgery: A Randomized Controlled Trial
Brief Title: Effect of ORI-guided Oxygen Titration on Oxidative Stress in Rhinoplasty Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Recep Karakaşoğlu, MD, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DLKCH-AR-RK-01
Record Dates: First submitted 2025-08-21; First posted 2025-09-05 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Rhinoplasty; Oxidative Stress; Hyperoxia; Oxygen Reserve Index
Keywords: Rhinoplasty surgery; Oxygen Reserve Index; Oxidative Stress; Hyperoxia
MeSH Terms: conditions — Hyperoxia

STUDY DESIGN:
Intervention Model Description: On the day of surgery, patients were randomly assigned into two groups -ORI group (Group R) and control group (Group C)- using the sealed envelope method. Patients in Group R received ORI monitoring in addition to intraoperative standart monitoring (ECG, pulse oximetry, non-invasive arterial blood pressure). For this purpose, an ORI sensor (RD Rainbow SET sensor, Masimo Corp., Irvine, CA, USA) was placed on the fourth finger of the upper extremity where there was no blood pressure cuff. The sensor was wrapped to prevent exposure to light and connected to an oximeter device (Raical-7® Pulse CO-Oximater®, Masimo Corp., Irvine, CA, USA). Patients in Group C received only standard monitoring.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both the clinicians involved in intraoperative patient management and the researchers responsible for data collection were blinded to group assignments. Additionally, randomization was performed on the day of surgery using the sealed envelope method, whereby patients were randomly assigned to either the ORI group (Group R) or the control group (Group C).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ORI group (Group R) (Active Comparator): Patients in Group R received ORI monitoring in addition to intraoperative standart monitoring (ECG, pulse oximetry, non-invasive arterial blood pressure). For this purpose, an ORI sensor (RD Rainbow SET sensor, Masimo Corp., Irvine, CA, USA) was placed on the fourth finger of the upper extremity where there was no blood pressure cuff. The sensor was wrapped to prevent exposure to light and connected to an oximeter device (Raical-7® Pulse CO-Oximater®, Masimo Corp., Irvine, CA, USA).In Group R, mask ventilation was administered with 50% oxygen. FiO₂ was titrated between 30% and 50% under the guidance of ORI and SpO₂ values. Accordingly, if SpO₂ was ≥ 98%, FiO₂ was reduced in 5% increments to a minimum of 30%, aiming to achieve an ORI value of 0 or as close to 0 as possible.
  Interventions: Device: FiO₂ titration, under the guidance of ORI
- Control group (Group C) (Active Comparator): Patients in Group C received only standard monitoring. Mask ventilation was administered with 100% oxygen. FiO₂ was maintained at 50% throughout the surgery, provided that SpO₂ remained ≥ 98%.
  Interventions: Device: Conventional oxygen administration

INTERVENTIONS:
Device: FiO₂ titration, under the guidance of ORI — In Group R, FiO₂ was titrated between 30% and 50% under the guidance of ORI and SpO₂ values. Accordingly, if SpO₂ was ≥ 98%, FiO₂ was reduced in 5% increments to a minimum of 30%, aiming to achieve an ORI value of 0 or as close to 0 as possible.
  Arms: ORI group (Group R)
Device: Conventional oxygen administration — In Group C, FiO₂ was maintained at 50% throughout the surgery, provided that SpO₂ remained ≥ 98%.
  Arms: Control group (Group C)

SUMMARY:
The aim of this study is to evaluate whether the use of Oxygen Reserve Index (ORİ) can prevent hyperoxia in patients undergoing rhinoplasty surgery and whether it can reduce oxidative stress caused by hyperoxia.

DETAILED DESCRIPTION:
ORI is a continuous, non-invasive parameter provided by new-generation pulse oximeters utilizing multi-wavelength pulse oximetry technology. ORI serves as an important monitoring tool for detecting both hyperoxemia and desaturation in patients with decreased PaO₂ levels. Studies have demonstrated that ORI provides values within a range of 0 to 1, and an ORI value of 0 corresponds to a PaO₂ level between 80 and 125 mmHg.

Oxygen is commonly used in clinical practice to prevent or treat hypoxia; however, excessive use may lead to oxidative stress. Oxidative stress is defined as a disruption of the oxidative balance resulting from an increased generation of reactive oxygen species (ROS) during cellular metabolism and an insufficient level of antioxidants to detoxify them. ROS are formed by the reaction of molecular oxygen with H₂O, the most stable form of oxygen. In this reaction, the stepwise addition of electrons to molecular oxygen (O₂) leads to the formation of superoxide anion (O₂ˉ), hydrogen peroxide (H₂O₂), and hydroxyl radical (-OH). Among these, the hydroxyl radical is the most reactive form of oxygen radicals.

Although ROS are essential for normal cellular functions such as intracellular signaling and defense against external threats, their excessive production can lead to molecular and cellular dysfunction. Excessive ROS attack nucleotide bases in nucleic acids, amino acid side chains in proteins, and double bonds in unsaturated fatty acids, resulting in oxidative stress that damages DNA, RNA, proteins, and lipids, leading to structural and metabolic changes in cells.

The primary aim of the investigators in this study is to determine whether ORI-guided oxygen titration during rhinoplasty surgery can help prevent hyperoxia and reduce oxidative stress compared with conventional oxygen therapy. To evaluate oxidative stress, thiol-disulfide balance and ischemia-modified albumin (IMA) levels will be assessed in the participants.

ELIGIBILITY:
Inclusion Criteria:

* classified as ASA physical status I or II

Exclusion Criteria:

* under 18 years of age
* ASA classification greater than II
* Mallampati score of 3 or 4
* findings suggestive of difficult intubation during physical examination
* any pathological findings on chest X-ray evaluation (e.g., pleural effusion, nodular density increase, emphysema, atelectasis, calcification, mediastinal widening, or infiltration)
* a history of circulatory disorders
* hematocrit or hemoglobin values outside the normal range (Hemoglobin: 12-16 g/dL for males, 11-14 g/dL for females; Hematocrit: 36-48% for males, 33-42% for females)
* a known hypersensitivity to any anesthetic agent to be used in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Change in thiol-disulfide balance. | preoperative to end of surgery (before awakening)
  Plasma native thiol, total thiol, and disulfide levels will be measured. The disulfide-to-thiol ratio will be used as a marker of oxidative stress. Unit of Measure: µmol/L
Change in ischemia-modified albumin (IMA) levels. | preoperative-end of surgery (before awakening)
  Serum IMA levels will be measured as an indicator of oxidative stress. IMA reflects modification of the N-terminal region of albumin by reactive oxygen species (ROS). Unit of Measure: Absorbance Units (ABS units)

SECONDARY OUTCOMES:
PaO₂ levels. | From baseline (after intubation) to end of surgery (before awakening)
  To compare intraoperative PaO₂ changes between ORI and Control groups. Arterial blood gas samples were obtained from all patients after intubation, at the 2nd hour of surgery, and at the end of the procedure before awakening.

CONTACTS AND LOCATIONS:
Overall Officials: Banu E Çevik, MD, Study Director — University of Health Sciences, Kartal Dr. Lütfi Kırdar City Hospital; Fatih D Geyik, MD, Principal Investigator — University of Health Sciences, Kartal Dr. Lütfi Kırdar City Hospital; Kemal T Saraçoğlu, MD, Principal Investigator — University of Health Sciences, Kartal Dr. Lütfi Kırdar City Hospital; Recep karakaşoğlu, MD, Principal Investigator — University of Health Sciences, Kartal Dr. Lütfi Kırdar City Hospital
Locations (1):
- Kartal Dr. Lütfi Kırdar City Hospital, Istanbul, kartal, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karakasoglu R, Geyik FD, Cevik BE, Saracoglu KT. The effect of oxygen reserve index guided oxygen titration on oxidative stress in rhinoplasty surgery: a randomized controlled trial. BMC Anesthesiol. 2025 Nov 4;25(1):542. doi: 10.1186/s12871-025-03424-0. PMID 41188744